CLINICAL TRIAL: NCT00058188
Title: A Phase III Randomized Study of Zolendronate Bisphosphonate Therapy for the Prevention of Bone Loss in Men With Prostate Cancer Receiving Long-Term Androgen Deprivation
Brief Title: Zolendronate for the Prevention of Bone Loss in Men w/ Prostate CA on Long-Term Androgen Deprivation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed by the research committee
Sponsor: Northwestern University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NU 02U1
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-10

CONDITIONS: Osteoporosis; Prostate Cancer
Keywords: osteoporosis; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Osteoporosis; Prostatic Neoplasms | interventions — Cholecalciferol; Calcium Gluconate; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive zoledronate IV over 15 minutes on day 1 and oral calcium gluconate and oral cholecalciferol daily. Courses repeat every 3 months for 12 months in the absence of toxicity.
  Interventions: Dietary Supplement: cholecalciferol; Drug: calcium gluconate; Drug: zoledronic acid
- Arm II (Active Comparator): Patients receive oral calcium gluconate and oral cholecalciferol as in arm I.
  Interventions: Dietary Supplement: cholecalciferol; Drug: calcium gluconate

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Given orally
Drug: calcium gluconate — Given orally
Drug: zoledronic acid — Given IV
  Arms: Arm I

SUMMARY:
RATIONALE: Zoledronate may prevent bone loss associated with long term androgen deprivation therapy. It is not yet known whether zoledronate combined with calcium is more effective than calcium alone in preventing bone loss.

PURPOSE: Randomized phase III trial to compare the effectiveness of zoledronate combined with calcium with that of calcium alone in preventing bone loss in patients with stage III or stage IV prostate cancer who have received long-term androgen deprivation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare bone loss in patients receiving long-term androgen deprivation therapy for stage III or IV prostate cancer when treated with supportive care with vs without zoledronate.
* Compare the percentage change in lumbar spine and hip bone density in patients treated with these regimens.
* Compare markers of bone formation and resorption in patients treated with these regimens.
* Compare the incidence of skeletal events (pathologic and non-pathologic bone fractures, spinal cord compression, surgery to bone, and radiotherapy to bone) in patients treated with these regimens.
* Compare the incidence of new or progressive bone metastatic disease in patients treated with these regimens.
* Compare the survival rate of patients treated with these regimens.

OUTLINE: Patients are stratified according to race (black vs other). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive zoledronate IV over 15 minutes on day 1 and oral calcium gluconate and oral cholecalciferol daily. Courses repeat every 3 months for 12 months in the absence of toxicity.
* Arm II: Patients receive oral calcium gluconate and oral cholecalciferol as in arm I.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 72 patients (36 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * Stage III or IV disease
* Received at least 3 months of prior androgen deprivation therapy (no maximum amount/time) by either surgical or medical castration

  * Medical castration may be by intermittent or continuous androgen suppression via single- or combined-drug androgen blockade
* Continued concurrent androgen deprivation therapy required throughout study participation
* No bone metastases by baseline bone scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 1 year

Hematopoietic

* Not specified

Hepatic

* Bilirubin less than 3 times upper limit of normal (ULN)
* AST and ALT less than 3 times ULN
* No chronic liver disease

Renal

* Creatinine no greater than 2.0 mg/dL

Other

* Fertile patients must use effective contraception
* No Paget's disease
* No Cushing's disease
* No hyperthyroidism
* No hyperprolactinemia

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior chemotherapy for prostate cancer allowed

Endocrine therapy

* See Disease Characteristics
* More than 12 months since prior suppressive doses of thyroxine or calcitonin
* More than 6 months since prior corticosteroids
* Concurrent corticosteroids allowed (after enrollment on study)

Radiotherapy

* Prior radiotherapy for prostate cancer allowed

Surgery

* See Disease Characteristics

Other

* More than 12 months since prior bisphosphonate therapy (oral or IV)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Bennett, MD, PhD, Study Chair — Robert H. Lurie Cancer Center
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - John H. Stroger Hospital of Cook County, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PIs departure from the institution was sudden and due unforeseen serious circumstances. Due to this, no data was collected for this study nor can be reported on.
Groups:
- Treatment With Zoledronate, Calcium and Cholecalciferol: Patients receive zoledronate IV over 15 minutes on day 1 and oral calcium gluconate and oral cholecalciferol daily. Courses repeat every 3 months for 12 months in the absence of toxicity.
  cholecalciferol: Given orally
  calcium gluconate: Given orally
  zoledronic acid: Given IV
- Treatment With Calcium and Cholecalciferol: Patients receive oral calcium gluconate and oral cholecalciferol as in arm I.
  cholecalciferol: Given orally
  calcium gluconate: Given orally
Period: Overall Study
Arm/Group | Treatment With Zoledronate, Calcium and Cholecalciferol | Treatment With Calcium and Cholecalciferol
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to the unique situation of the PI, no data was collected for this study nor can be reported on.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Zoledronate, Calcium and Cholecalciferol | Treatment With Calcium and Cholecalciferol | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Bone Density Change as Measured by Dual-energy X-ray Absorptiometry From Baseline to 13 Months
Description: To assess bone density change as measured by dual-energy x-ray absorptiometry
Time Frame: Bone scan taken at baseline and month 13
Population: Due to the unique situation of the PI, no data was collected for this study nor can be reported on.
Arm/Group | Treatment With Zoledronate, Calcium and Cholecalciferol | Treatment With Calcium and Cholecalciferol
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage Change in Lumbar Spine and Hip Bone Density as Measured by Plain Film X-rays of Lumbar Spine and Pelvis From Baseline to 13 Months
Description: To assess the percentage change in lumbar spine and hip bone density as measured by plain film x-rays of lumbar spine and pelvis
Time Frame: Lumbar spine and hip bone density taken at baseline and month 13.
Population: Due to the unique situation of the PI, no data was collected for this study nor can be reported on.
Arm/Group | Treatment With Zoledronate, Calcium and Cholecalciferol | Treatment With Calcium and Cholecalciferol
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Markers of Bone Formation and Resorption
Description: To assess markers of bone formation and resorption.
Time Frame: Bone alkaline phosphatase taken at baseline, month 6 and month 13.
Population: Due to the unique situation of the PI, no data was collected for this study nor can be reported on.
Arm/Group | Treatment With Zoledronate, Calcium and Cholecalciferol | Treatment With Calcium and Cholecalciferol
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Skeletal Events (Pathologic and Non-pathologic Bone Fractures, Spinal Cord Compression, Surgery to Bone, and Radiotherapy to Bone)
Description: To assess the incidence of skeletal events (pathologic and non-pathologic bone fractures, spinal cord compression, surgery to bone, and radiotherapy to bone)
Time Frame: PSA taken at baseline, month 3, month 6, month 9, month 12 and month 13. CT scan of abdomen and pelvis taken at baseline and month 13. Serum testosterone, estradiol, parathyroid taken at baseline, month 6 and month 13.
Population: Due to the unique situation of the PI, no data was collected for this study nor can be reported on.
Arm/Group | Treatment With Zoledronate, Calcium and Cholecalciferol | Treatment With Calcium and Cholecalciferol
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of New or Progressive Bone Metastatic Disease
Description: To assess the incidence of new or progressive bone metastatic disease
Time Frame: Serum osteocalcin and serum bone alkaline phosphatase taken at baseline, month 6 and month 13.
Population: Due to the unique situation of the PI, no data was collected for this study nor can be reported on.
Arm/Group | Treatment With Zoledronate, Calcium and Cholecalciferol | Treatment With Calcium and Cholecalciferol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events timeframe is not known. There is no data for this study.
Description: Due to the unique situation of the PI, no data was collected for this study nor can be reported on.
Arm/Group | Treatment With Zoledronate, Calcium and Cholecalciferol | Treatment With Calcium and Cholecalciferol
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No